CLINICAL TRIAL: NCT03790761
Title: Guam Healthy Relationships Education Program
Acronym: GHREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WestCare Pacific Islands, Inc. (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5589
Record Dates: First submitted 2018-11-14; First posted 2019-01-02 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Health Behavior
Keywords: Guam; healthy relationships; non-profit organization; PREP 8.0 curriculum
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PREP 8.0 Curriculum (Experimental): All participants enrolled in the program will be given the PREP 8.0 curriculum - there will be no comparison group.
  Interventions: Behavioral: PREP 8.0 Curriculum

INTERVENTIONS:
Behavioral: PREP 8.0 Curriculum — The PREP 8.0 curriculum is an experiential curriculum designed to be implemented in a workshop or educational setting. Using techniques of cognitive-behavioral marital therapy and communication-oriented marital enhancement, PREP aims to help couples achieve high levels of relationship functioning and prevent marital problems. The PREP approach is based on research in the field of relational and marital health and success conducted at the University of Denver.

SUMMARY:
The Guam Healthy Marriage Partnership (GHMP), a comprehensive culturally responsive program that will foster healthy relationships and marriages on the island of Guam.

DETAILED DESCRIPTION:
The proposed Guam Healthy Relationships Education Program will improve the quality of life for individuals/couples in Guam by using culturally responsive approaches to foster healthy relationships and marriages using an Observational approach as there will be no comparison group, only the control group. Project activities include a 6-month education program of interactive curriculum-based groups and positive social/recreational activities to achieve positive outcomes for individuals/couples, community awareness events, and community and parenting skills training. The services offered is entrenched in cultures and traditions that are meaningful to the people of Guam, and includes capacity building and community awareness activities that will change community, family, and peer normative environments and attitudes.

ELIGIBILITY:
Inclusion Criteria:

* Currently in a long-term relationship, does not have to include marriage
* Must be at least 18 years old
* At least one of the partners need to be between the ages of 18-35 years old

Exclusion Criteria:

* Under the age of 18 years
* Not in a long-term relationship

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 556 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Relationship Satisfaction | The pre-test is administered before starting the curriculum and the post-test is administered immediately following the conclusion of the curriculum.
  The PREP 8.0 curriculum pre- and post-test will be administered to program participants to determine if there are any changes in relationship satisfaction.

SECONDARY OUTCOMES:
Change in Intimate Partner Violence | The screening is administered before starting the curriculum and the screening is administered again immediately following the conclusion of the curriculum.
  The HITS Screening Assessment will be administered to program participants to determine if there are any changes in intimate partner violence as a result of participating in the PREP 8.0 curriculum.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Rhea, Ed.D., Principal Investigator — WestCare Foundation, Inc.
Locations (1):
- WestCare Pacific Islands Reflection Center, Hagåtña, Guam

IPD SHARING:
Plan to Share IPD: Undecided
WestCare is willing to work with other researchers in the field for the betterment of the quality of life of Guam's community. An individual participant data (IPD) will be determined based upon potential partner.